CLINICAL TRIAL: NCT06847984
Title: Antimicrobial Effect of Curcumin on Oral Microbiome Versus Chlorohexidine in High Caries Risk Individuals
Brief Title: Antimicrobial Effect of Curcumin Versus Chlorohexidine on Oral Microbiome
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Salma Basyouni, Dr, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Curc-Chlorohexidine
Record Dates: First submitted 2025-02-16; First posted 2025-02-26 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Dental Caries; Dental Plaque Index; Oral Microbiome
Keywords: oral microbiome, curcumin, chlorohexidine, antimicrobial
MeSH Terms: conditions — Dental Caries | interventions — Curcumin

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: statistician
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- chlorohexidine (Active Comparator): Participants were instructed to rinse with 10 mL of mouthwash for
  1 minute, once daily for 1 week of each month. This regimen was repeated monthly for a period of 1 year
  Interventions: Other: Chlorohexidine
- curcumin (Experimental): Participants were instructed to rinse with 10 mL of mouthwash for
  1 minute, once daily for 1 week of each month. This regimen was repeated monthly for a period of 1 year
  Interventions: Dietary Supplement: Curcumin

INTERVENTIONS:
Dietary Supplement: Curcumin — Participants were instructed to rinse with 10 mL of mouthwash for
  1 minute, once daily for 1 week of each month. This regimen will be repeated monthly for a period of 1 year.
  Arms: curcumin
Other: Chlorohexidine — Participants were instructed to rinse with 10 mL of mouthwash for 1 minute, once daily for 1 week of each month. This regimen will be repeated monthly for a period of 1 year
  Arms: chlorohexidine

SUMMARY:
Dental caries, one of the world's most common infectious diseases, is a biofilm-mediated, sugar-driven, dynamic disease. It has an impact on physical, mental, and social health and is extremely costly to society. It is a complex disease with microbiological, behavioral, genetic, and environmental components. Recently, it has been demonstrated in the literature that the development of dental caries is strongly related with the microbiota in the oral cavity. So, a detailed understanding of caries microbiology is needed.

Oral microbiome, oral microbiota or oral microflora refers to the microorganisms found in the human oral cavity that was first identified by the Dutchman Antony van Leeuwenhoek using a microscope constructed by him. In 1674, he observed his own dental plaque and reported "little living animalcules prettily moving".

Human microbiome consists of a core microbiome which is common to all the individuals and a variable microbiome that is unique to individuals depending on the lifestyle and physiological differences. Dental caries, as a process determined by lifestyle, may be subject to activation in each period of human life if hygiene and diet are neglected even for a period as short as a few weeks.

Previous hypotheses suggest that Streptococcus mutans is the primary pathogen in the development of dental caries in both children and adults. However, recently published papers provide a partially different perspective on the role of bacteria in the caries process, known as the "extended caries ecological hypothesis," which attempts to demonstrate that the role of S. mutans in the initiation of dental caries may not be as dominant as previously assumed, but there is agreement that they have the highest cariogenic potential.

It is now believed that the disease is caused by microorganisms belonging to the natural flora of the oral cavity: the oral microbiome. There is a dynamic equilibrium between microorganisms as well as between the micro flora and the 7 host, and the disease develops as a result of a microbiological imbalance within the biofilm.

Therefore, a better understanding of processes of oral biofilm formation and function is necessary to the development of novel, successful, rational approach for antimicrobial strategies and caries prevention and treatment.

Primary caries can be prevented, stopped and treated by regular plaque removal and remineralization mechanisms. Fluorides play a central role in the prevention of dental caries and are being used extensively and therapeutically for the inactivation of incipient carious lesions. However, regarding the high cost of dental clinic setting and difficult access to the oral health care service that is not well-covered in certain countries; the treatment strategy should move towards the preventive, simple, accessible, less costly methods.

The frequent use and abuse of the currently used therapeutic agents has led to the evolution of resistant strains of common pathogens as well as increased incidence of adverse effects associated with their usage. Therefore, natural phytochemicals extracted from plants used as traditional medicines are therefore seen as a good alternative source.

Pharmaceutical plants have been used throughout human history to treat a variety of diseases. According to the World Health Organization, almost 80% of the world's population relies on traditional medicinal plants for primary health care. In dentistry, there is a growing need to develop natural materials with anti-caries qualities.

Curcumin (CUR), a dietary natural product extracted from the root of turmeric (the major constituent of Curcuma longa L. or turmeric), which is widely used as a flavoring and coloring agent has many pharmacological activities including anti-inflammatory and antitumor properties. In addition, CUR has been shown to have anti-bacterial, whitening, and antioxidative activities. Various studies on widespread Polyphenolic compounds suggest that curcumin inhibits the bacterial effect by reducing the production of acid and stopping the adherence of bacteria to the tooth surface. Song et al. found that curcumin could significantly inhibit the adhesiveness of S. mutans by its effects on collagen and fibronectin. The antibacterial action of curcumin involves the disruption of the bacterial membrane, inhibition of the production of bacterial virulence factors and biofilm formation, and the induction of oxidative stress. These characteristics also contribute to explain how curcumin acts a broad-spectrum antibacterial adjuvant. So, the aim of the following interventional study is to evaluate the effect of curcumin on oral microbiome obtained from salivary samples of high caries risk patients in vitro and assess the antiplaque and anticariogenic effect of curcumin mouth wash in high caries risk patients in a randomized controlled clinical trial compared to chlorohexidine mouth wash.

ELIGIBILITY:
Inclusion Criteria:

* Provide informed consent.
* Patients accept the one-year follow-up period.
* Cooperative patients.
* The study recruited volunteers of both genders
* Age from 21 to 45 years
* Patients classified at high risk of caries

Exclusion Criteria:

* Patients undergoing orthodontic treatment.
* Periodontal compromised patients.
* Smokers.
* Pregnant women.
* Patients with physical or mental disability
* Patient with removable prosthesis

Ages: 21 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 54 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Caries incidence | Baseline, 7, 30 days, 3 months, 1 year
  caries incidence will be checked using DMF (Decayed, Missing or Filled Surfaces,)

SECONDARY OUTCOMES:
Plaque | Baseline, 7, 30 days, 3 months, 1 year
  plaque will be checked using plaque index. minimal value (0): absence of microbial plaque. maximum value (3): large amount of plaque in sulcus or pocket along the free gingival margin Higher scores mean a worse outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
still undecided,

REFERENCES:
- See also: Caries Preventive and Antibacterial Effects of Two Natural Mouthwashes vs Chlorhexidine in High Caries-risk Patients: A Randomized Clinical Trial — https://www.google.com.eg/search?q=+Caries+Preventive+and+Antibacterial+Effects+of+Two+Natural+Mouthwashes+vs%0D%0A+Chlorhexidine+in+High+Caries-risk+Patients%3A+A+Randomized+Clinical+Trial&sca_esv=54fcc75b4f72cd60&source=hp&ei=voyuZ8vdA_OekdUP0NDuyAY&iflsig=ACkRmUkAAAAAZ66azsvNgGBw7zVNyA5kiOD6T-g1Bxyl&ved=0ahUKEwjLtLzY8sGLAxVzT6QEHVCoG2kQ4dUDCBc&uact=5&oq=+Caries+Preventive+and+Antibacterial+Effects+of+Two+Natural+Mouthwashes+vs%0D%0A+Chlorhexidine+in+High+Caries-risk+Patients%3A+A+Randomized+Clinical+Trial&gs_lp=Egdnd3Mtd2l6IpMBIENhcmllcyBQcmV2ZW50aXZlIGFuZCBBbnRpYmFjdGVyaWFsIEVmZmVjdHMgb2YgVHdvIE5hdHVyYWwgTW91dGh3YXNoZXMgdnMKIENobG9yaGV4aWRpbmUgaW4gSGlnaCBDYXJpZXMtcmlzayBQYXRpZW50czogQSBSYW5kb21pemVkIENsaW5pY2FsIFRyaWFsSABQAFgAcAB4AJABAJgBAKABAKoBALgBA8gBAPgBAvgBAZgCAKACAJgDAJIHAKAHAA&sclient=gws-wiz&sei=w4yuZ4utF9zc7_UP3YbIuAM